CLINICAL TRIAL: NCT01296841
Title: A Randomized Controlled Pilot: Use of Telemedicine To Provide Inflammatory Bowel Disease Outpatient Care
Brief Title: Telemedicine To Provide Inflammatory Bowel Disease Outpatient Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Soetikno, Clinical Professor, Chief of Endoscopy, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TELEMED PA
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
Keywords: telemedicine; remote consultation; telehealth; ehealth; image archiving; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard encounter (No Intervention): Standard "in-house" clinical visit between patient and physician.
- Telemedicine Encounter (Experimental): Remote clinical appointment between patient and physician.
  Interventions: Device: Collaborative Imaging

INTERVENTIONS:
Device: Collaborative Imaging — Hardware and software communication tools to provide clinical care from a distance.
  Other Names: Telemedicine
  Arms: Telemedicine Encounter

SUMMARY:
The investigators hypothesize that outpatient clinical care of Inflammatory Bowel Disease patients may be provided using a new computerized system over standard network - called Collaborative Imaging - with similar patient experience compared to a conventional clinic visit.

DETAILED DESCRIPTION:
Significant advances in gastroenterology have led the field to grow into a number of advanced subspecialties: inflammatory bowel disease (IBD), motility, therapeutic endoscopy, and transplant hepatology. Telemedicine, the application of information technology in support of health care delivery from a distance, has been employed with good success in various chronic conditions with excellent patient satisfaction.

Primary Aim: Our primary study endpoint was measuring patient clinical experience between two groups: A telemedicine remote clinic visit and a standard "in-house" visit.

Secondary Aim: To compare standard clinic metrics including clinic wait time, patient throughput, and appointment time between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old) outpatient IBD patients in the Veterans Affairs medical system

Exclusion Criteria:

* VA patients without IBD
* Hospitalized IBD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Kaltenbach, MD MS, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- Veterans Affairs Palo Alto, Palo Alto, California, United States

REFERENCES:
- [Background] Telleman H, Burger TF, Mulder CJ. Evolution of gastroenterology training. World J Gastroenterol. 2009 Apr 21;15(15):1793-8. doi: 10.3748/wjg.15.1793. PMID 19370773
- [Background] Fisher ES, Welch HG. The future of the Department of Veterans Affairs health care system. JAMA. 1995 Feb 22;273(8):651-5. No abstract available. PMID 7844876
- [Background] Dorsey ER, Deuel LM, Voss TS, Finnigan K, George BP, Eason S, Miller D, Reminick JI, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Biglan KM. Increasing access to specialty care: a pilot, randomized controlled trial of telemedicine for Parkinson's disease. Mov Disord. 2010 Aug 15;25(11):1652-9. doi: 10.1002/mds.23145. PMID 20533449
- [Background] Verhoeven F, Tanja-Dijkstra K, Nijland N, Eysenbach G, van Gemert-Pijnen L. Asynchronous and synchronous teleconsultation for diabetes care: a systematic literature review. J Diabetes Sci Technol. 2010 May 1;4(3):666-84. doi: 10.1177/193229681000400323. PMID 20513335
- [Background] Grogan-Johnson S, Alvares R, Rowan L, Creaghead N. A pilot study comparing the effectiveness of speech language therapy provided by telemedicine with conventional on-site therapy. J Telemed Telecare. 2010;16(3):134-9. doi: 10.1258/jtt.2009.090608. Epub 2010 Mar 2. PMID 20197354
- [Background] van der Heijden JP, Spuls PI, Voorbraak FP, de Keizer NF, Witkamp L, Bos JD. Tertiary teledermatology: a systematic review. Telemed J E Health. 2010 Jan-Feb;16(1):56-62. doi: 10.1089/tmj.2009.0020. PMID 20064068
- [Background] Wallace P, Haines A, Harrison R, Barber JA, Thompson S, Roberts J, Jacklin PB, Lewis L, Wainwright P; Virtual Outreach Project Group. Design and performance of a multi-centre randomised controlled trial and economic evaluation of joint tele-consultations [ISRCTN54264250]. BMC Fam Pract. 2002 Jan 11;3:1. doi: 10.1186/1471-2296-3-1. Epub 2002 Jan 11. PMID 11835692
- See also: telemedicine personal computer — http://www.apple.com/imac/
- See also: telemedicine personal computer — http://www.apple.com/macpro/
- See also: telemedicine headset — http://www.plantronics.com/north_america/en_US/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Encounter | Telemedicine Encounter
Started | 19 | 15
Completed | 19 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Encounter | Telemedicine Encounter | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 24
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.6) | 62.8 (11.5) | 60.4 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Patient Clinical Experience
Description: We used a validated Ware Specific Visit Questionnaire to assess patients' satisfaction with their clinic-visit encounter. This is a 14-item questionnaire on doctor-patient interaction including factors such as attention to complaints, technical skills, and personal manner (courtesy,and ease of appointment scheduling and is based on a five-point Likert scale (1 excellent to 5 poor). Patients completed the questionnaire at the time of the visit. The 14 item scores were individually scored and then averaged to provide the final overall value.
Time Frame: Clinic Visit
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telemedicine: clinic experience (mean ± SD, 1 excellent, 5 poor)
- Standard: clinic experience (mean±SD)
Arm/Group | Telemedicine | Standard
Number analyzed (Participants) | 15 | 19
units on a scale | 1.2 (0.4) | 1.3 (0.5)
Statistical Analysis 1: Comparison: Telemedicine vs Standard; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; We performed t-test statistics for univariate comparisons for continuous variables

2. Secondary Outcome: Clinic Appointment Duration
Description: The investigators recorded appointment duration in minutes.
Time Frame: Clinic Visit
Population: Pilot.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard Encounter | Telemedicine Encounter
Number analyzed (Participants) | 19 | 15
Minutes | 59 (18) | 60 (25)

3. Secondary Outcome: Clinic Appointment Wait Time
Description: The investigators recorded clinic appointment wait time duration in minutes
Time Frame: Clinic Visit
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Encounter | Telemedicine Encounter
Number analyzed (Participants) | 19 | 15
minutes | 18 (14.5) | 25 (25)

ADVERSE EVENTS:
Arm/Group | Standard Encounter | Telemedicine Encounter
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes